CLINICAL TRIAL: NCT06954610
Title: CARE-AF: Cardiac Assessment for Recurrent Stroke Risk Evaluation in Atrial Fibrillation
Brief Title: Cardiac Assessment for Recurrent Stroke Risk Evaluation in Atrial Fibrillation
Acronym: CARE-AF
Status: Recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: STD0007325
Record Dates: First submitted 2025-04-16; First posted 2025-05-01 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Ischemic Stroke; Atrial Fibrillation; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Vascular Diseases; Arrhythmias, Cardiac; Heart Diseases; Brain Infarction; Brain Ischemia; Infarction Cerebral; Stroke; Cardioembolic Stroke; Ischemia
Keywords: Ischemic stroke; Direct oral anticoagulation; Anticoagulation; Breakthrough stroke; Risk stratification; Atrial fibrillation; Anticoagulant therapy; Direct oral anticoagulant
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Vascular Diseases; Arrhythmias, Cardiac; Heart Diseases; Brain Infarction; Brain Ischemia; Cerebral Infarction; Stroke; Embolic Stroke; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Background

Atrial fibrillation (AF) is the most common cardiac arrhythmia, affecting up to 10% of the elderly. Ischemic stroke is the main complication of AF and cardioembolism is one of the leading causes of ischemic stroke, accounting for approximately one third of cases. Oral anticoagulant therapy (OAC) is a cornerstone in stroke prevention in patients with AF. According to randomized controlled trials of direct oral anticoagulants, a residual risk of ischemic stroke of 1-2% per year for so-called "breakthrough stroke" remains, despite adequate intake of OAC. The majority (>70%) of these breakthrough strokes are cardioembolic in nature and only a minority are related to medication issues (e.g. non-compliance) or other, non-AF related etiologies. Stroke recurrence risk after such a breakthrough stroke markedly increases to 8-9% per year indicating a particularly high-risk situation. Why OAC fails in certain patients, but not in others remains as poorly understood, as does the reason why the subsequent risk of stroke is so high.

Current risk stratification tools, such as the widely used CHA2DS2-VA(Sc)-score, fail to predict stroke risk in such a high-risk cohort, as they were intended to guide the initiation of OAC in low to moderate risk patients. In light of new therapeutic strategies currently being investigated, such as percutaneous left atrial appendage occlusion in patients with breakthrough strokes (ELAPSE - NCT05976685) or in AF-patients deemed high-risk (LAAOS IV - NCT05963698), improved risk stratification and characterization of high-risk AF patients is highly warranted.

Several clinical factors, such as those reflected in the CHA2DS2-VA(Sc)-score, and especially a high AF-burden are associated with increased risk of cardioembolic stroke. Several cardiac serum biomarkers are thought to be surrogates not only of cardiac function, but also of cardioembolic risk. Reflecting ventricular and atrial wall tension, myocardial injury, oxidative stress and thrombogenicity, elevated NT-proBNP, MR-proANP, high-sensitive Troponin T and D-Dimers have all been associated with cardioembolic stroke in different AF and non-AF populations. As the main location of thrombus formation, the left atrium (LA) and more specifically its appendage (LAA) are of particular interest in the pathogenesis of cardioembolism. Pronounced LA-enlargement, compared to a normal-sized LA, correlates with an increased risk of cardioembolism in AF-patients. As over 80% of thrombi form within the LAA, several LAA-characteristics, such as slower LAA-flow velocity and larger LAA-orifice area have also been demonstrated to be associated with higher stroke risk. Although there is data on each one of these factors, they have only been investigated in low to moderate risk populations, such as AF-patients without prior stroke, OAC-naïve patients, or even within the general population as a whole. Their role in high-risk AF-patients and in breakthrough stroke is unknown.

Hypothesis

The investigators hypothesize that specific clinical factors, serum cardiac biomarkers and markers of LA- and LAA-morphology and function are associated with breakthrough stroke / OAC-failure and may improve risk stratification.

Methods

CARE-AF is a single-center, prospective cohort study conducted at the Stroke Center of the Inselspital, University Hospital Bern, Switzerland. Patients with an index ischemic stroke and AF (breakthrough and non-breakthrough cases) will be enrolled. The investigators will collect clinical data, serum cardiac biomarkers and echocardiographic indices of the LA and LAA. All patients will receive standardized annual follow-ups until the end of the study, defined as 12 months after the inclusion of the last participant. The primary endpoint is ischemic stroke or systemic embolism during follow-up. First, in a cross-sectional design, the study will assess the association between serum cardiac biomarkers and echocardiographic indices among patients with breakthrough vs. non-breakthrough stroke as index event, applying multivariate regression models. Second, the investigators will perform a longitudinal analysis assessing the association between the variables mentioned above and breakthrough stroke as index event with the primary endpoint, using multivariate Cox regression models. The study aims to enroll a minimum of 500 patients, which provides sufficient power to detect a clinically meaningful adjusted hazard ratio for recurrent stroke of 1.5 with 80% power at an alpha level of 5%.

Conclusion

The results of this project will enhance understanding of the role of specific clinical factors, cardiac serum biomarkers and echocardiographic indices in the residual risk of stroke in patients with AF on anticoagulation therapy. They may improve current risk stratification and have the potential to help guide therapeutic decisions in high-risk situations considering evolving therapeutic possibilities.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Written informed consent (by patient, next of kin or legally authorised representative)
* Permanent, persistent, or paroxysmal AF previously known or diagnosed during the index hospitalisation
* Acute (≤7 days), symptomatic ischemic stroke

Exclusion Criteria:

* Life expectancy <1 year according to the opinion of the investigator
* Patient is unlikely to attend follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with ischemic stroke and atrial fibrillation that are admitted to the stroke center of the Inselspital, University Hospital Bern, Switzerland.
  Atrial fibrillation may be known prior to the index stroke or newly diagnosed and patients may be anticoagulated or not.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-11-04 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite of recurrent ischemic stroke or systemic embolism | Assessed in first follow-up visit at 12 months (+/- 30 days) after enrolment. Subsequent assessments/visits will be every 12 months and at the end of study (if last visit has taken place >90days prior). Minimal Follow up per patient is 12 months.
  * Ischemic stroke defined as new neurological symptoms lasting >24h and/or evidence of new ischemic lesions in neuroimaging (CT and/or MRI)
  * Systemic embolism, defined as an abrupt vascular insufficiency associated with radiological evidence of arterial occlusion of an extremity or internal organ, in absence of any other, more-likely etiology (e.g. trauma)
  * Will be assessed through structured telephone visits at every follow-up visit

SECONDARY OUTCOMES:
All-cause death | Assessed in first follow-up visit at 12 months (+/- 30 days) after enrolment. Subsequent assessments/visits will be every 12 months and at the end of study (if last visit has taken place >90days prior). Minimal Follow up per patient is 12 months.
  Death of all cause
  - Will be assessed through structured telephone visits at every follow-up visit
MACE (major adverse cardial events), defined as a composite outcome of myocardial infarction (MI), ischemic and haemorrhagic stroke, transient ischemic attack (TIA), systemic embolism and cardiovascular death | Assessed in first follow-up visit at 12 months (+/- 30 days) after enrolment. Subsequent assessments/visits will be every 12 months and at the end of study (if last visit has taken place >90days prior). Minimal Follow up per patient is 12 months.
  * Myocardial infarction, defined according to the 4th Universal Definition of MI as a combination of acute myocardial injury (changes in cardiac biomarkers) and evidence of acute myocardial ischemia derived from the clinical presentation, electrocardiographic changes, or the results of myocardial or coronary artery imaging.25
  * Transient ischemic attack, defined as a transient episode of neurologic dysfunction caused by focal ischemia (brain, spinal cord or retina) not fulfilling stroke-criteria
  * Intracranial haemorrhage, defined as intracranial haemorrhage (intraparenchymal, subarachnoid, sub-/epidural) not due to trauma
  * Cardiovascular death, resulting from cardio-/cerebrovascular causes (e.g. myocardial infarction, sudden cardiac or unwitnessed death, stroke etc.
  * Will be assessed through structured telephone visits at every follow-up visit
Episodes of symptomatic AF | Assessed in first follow-up visit at 12 months (+/- 30 days) after enrolment. Subsequent assessments/visits will be every 12 months and at the end of study (if last visit has taken place >90days prior). Minimal Follow up per patient is 12 months.
  Defined as symptoms attributable to AF that led to change in medication (initiation and/or change of rhythm and/or rate control medication), AF-ablation and / or electro-conversion.
  - Will be assessed through structured telephone visits at every follow-up visit
Functional outcome: modified Rankin Scale | Assessed in first follow-up visit at 12 months (+/- 30 days) after enrolment. Subsequent assessments/visits will be every 12 months and at the end of study (if last visit has taken place >90days prior). Minimal Follow up per patient is 12 months.
  Functional outcome measured using the modified Rankin Scale (mRS), ranging from 0 (no symptoms) to 6 (death)
  - Will be assessed through structured telephone visits at every follow-up visit
Functional outcome: Quality of life | Assessed in first follow-up visit at 12 months (+/- 30 days) after enrolment. Subsequent assessments/visits will be every 12 months and at the end of study (if last visit has taken place >90days prior). Minimal Follow up per patient is 12 months.
  Functional outcome measured as subjective quality of life with EQ5D-Score (EuroQol-5 dimensions score)
  * Assesses overall quality of life with a score ranging from 0 (worst) to 100 (best)
  * Assesses 5 dimensions of daily live, each ranging from 0 (no problem) to 5 (severe problem): Mobility, Self-Care, Activities of daily life, pain and discomfort, anxiety and depression
  * Will be assessed through structured telephone visits at every follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: David Seiffge, Prof. MD, Principal Investigator — Department of Neurology, Inselspital, University Hospital Bern, Switzerland
Locations (1):
- Inselspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No